CLINICAL TRIAL: NCT05353998
Title: Evaluating the Efficacy of Clinical Decision Support and Sleep Navigation to Enhance Primary to Specialty Care Management of Sleep Disordered Breathing
Brief Title: Efficacy of Clinical Decision Support and Sleep Navigation (Sleep PASS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-019762
Record Dates: First submitted 2022-03-15; First posted 2022-04-29 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Sleep-Disordered Breathing; Obstructive Sleep Apnea; Sleep
Keywords: Sleep Disordered Breathing; Sleep PASS
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Compact Disks

STUDY DESIGN:
Intervention Model Description: Caregiver-child dyads with a child who meets criteria for further SDB evaluation will be randomly assigned (1:1) to either the intervention condition, which is the CDS and the Sleep Navigation program, or to a CDS only condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Navigation group (Experimental): Caregiver-child dyads in this study arm (intervention condition) will participate in the Sleep Navigation program.
  Interventions: Other: CDS with Sleep Navigation
- CDS-only group (Other): Caregiver-child dyads in this study arm (control group) will not participate in the Sleep Navigation program, but will be directed to follow up with their primary care clinician as needed.
  Interventions: Other: CDS-only

INTERVENTIONS:
Other: CDS with Sleep Navigation — The Sleep Navigation program will involve 1-3 meetings between the Sleep Navigator (SN) and the participating family. Participants will also complete baseline and post-intervention assessments, and about 10 to 15 caregivers will be randomly invited to participate in an interview on the acceptability and feasibility of the program. The SN will provide: SDB and sleep health psychoeducation using Patient-Family Education handouts and videos that are currently part of usual care practices; Care coordination for scheduling of specialty care referral(s) for clinical SDB evaluation; Problem-solving for family-identified barriers to accessing specialty care; and Motivational interviewing to enhance family engagement, communication, and collaboration with the family's medical team.
  Arms: Sleep Navigation group
Other: CDS-only — Participants will complete baseline and post-intervention assessments. Participants will be able to follow-up with their primary care clinician as needed.
  Arms: CDS-only group

SUMMARY:
The purpose of the study is to examine the feasibility, acceptability, and initial outcomes of clinical decision support (CDS) and a Sleep Navigation program to enhance primary to specialty care management of pediatric sleep-disordered breathing (SDB).

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB), which ranges from mild snoring to severe obstructive sleep apnea, impacts up to 17% of all children and is a significant public health concern. Untreated SDB is associated with significant risks to child health and well-being, including child neurobehavioral problems, hypertension, and obesity. Despite the robust evidence base for treating SDB, there are notable racial, ethnic, and socioeconomic disparities in its prevalence and treatment; even when SDB is identified in primary care visits, referral rates to specialty care are extremely low.

This is a randomized controlled trial of the Sleep PASS program, with the primary objectives to (1) determine the feasibility and acceptability of CDS for SDB in primary care, and (2) determine the feasibility and acceptability of Sleep Navigation for patients with SDB who meet criteria for further clinical evaluation. The secondary objective is to examine the initial efficacy of CDS and Sleep Navigation on referral rates and rates of referral completion for SDB-related specialty care, caregiver SDB knowledge, and child sleep for patients with SDB who meet criteria for further clinical evaluation. Up to 200 caregiver-child dyads with a child (ages 2 years 0 months to < 18 years) who has been screened for SDB symptoms in Children's Hospital of Philadelphia primary care and meets criteria for further clinical evaluation will be recruited. Up to 70 primary care clinicians will also be recruited.

Eligible and interested caregiver-child dyads will be randomly assigned to the intervention condition (CDS with Sleep Navigation) or to the CDS only condition. The Sleep Navigation program will involve 1-3 meetings, conducted virtually, in-person, or via telephone, between the Sleep Navigator (SN) and the participating family. The SN will provide: SDB and sleep health psychoeducation using Patient-Family Education handouts and videos that are currently part of usual care practices; Care coordination for scheduling of specialty care referral(s) for clinical SDB evaluation; Problem-solving for family-identified barriers to accessing specialty care; and Motivational interviewing to enhance family engagement, communication, and collaboration with the family's medical team.

Study procedures involves medical record review, caregiver- and child-completed questionnaires, clinician-completed questionnaires, interviews, and Navigator sessions (for the Intervention condition). Following sleep screening as part of well child visit care, electronic health records and the sleep screener will be reviewed for eligibility. Eligible and interested participants will be scheduled for a baseline assessment visit that occurs in-person or electronically and includes informed consent (or e-consent), random assignment to the intervention condition (CDS with Sleep Navigation) or to the CDS only condition, and completion of baseline measures. The intervention group will start receiving the Sleep Navigation program 1-2 weeks following baseline assessment. The CDS only condition will be directed to follow up with their primary care clinician as needed. Post-intervention and follow-up assessment will occur within 8 months of baseline questionnaire completion. Clinicians will complete questionnaires at the post-intervention phase. Randomly selected caregiver-child dyads in the intervention condition and clinicians will be invited to participate in qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

Caregiver-child dyads:

1. Child is between 2 years and 17 years of age
2. Child has an abnormal SDB screen (i.e., a positive response to whether the child snores 3 or more nights/week) on the sleep screener used as part of well child visit care in the Children's Hospital of Philadelphia (CHOP) primary care network
3. Child receives well child care at Cobbs Creek or Karabots CHOP primary care network sites
4. Parental/guardian permission (informed consent) and if applicable, child assent
5. Caregiver participant is the parent or legal guardian of the child subject
6. Caregiver is 18 years of age or older
7. English-speaking

   Clinicians:
8. Primary care clinician practicing at Cobbs Creek or Karabots CHOP primary care network sites
9. English-speaking

Exclusion Criteria:

Caregiver-child dyads:

1. Caregiver is not the parent or legal guardian of child participant or is <18 years of age
2. Non-English speaking, as intervention sessions and qualitative interviews will be conducted in English
3. Child receives well child care at a non-participating primary care site at enrollment
4. Caregivers/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

   Clinicians:
5. Does not see patients at Cobs Creek or Karabots CHOP primary care network sites
6. Non-English speaking, as qualitative interviews will be conducted in English

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
CDS feasibility (proportion of patients screened for SDB at well child visits of all those eligible for screening at well child visits over the study period) | up to 12 months
  Proportion of patients screened for SDB at well child visits will be calculated with data from the electronic health records.
Clinician Decision Support Acceptability | up to 12 months
  Clinician Decision Support acceptability will be measured through clinician-completed system usability survey.
  This measure is rated on a 5-point Likert scale (1=strongly disagree; 2=somewhat disagree; 3=neither agree or disagree; 4=somewhat agree; and 5=strongly agree) with a range in score from 12 to 60. Higher total scores indicate better acceptability.
Acceptability of the CDS Tool | up to 12 months
  CDS acceptability will be measured by semi-structured qualitative interviews completed by the clinicians. Up to 15 primary care clinicians will be invited to participate in an interview focused on acceptability of the CDS tool. The interview includes multiple, open-ended questions completed by the clinician.
Sleep Navigator feasibility (number of Sleep Navigation activities completed among those randomized to receive Sleep Navigation) | within 8 months of baseline assessment
  Feasibility will be measured using data from the Sleep Navigator-completed intervention-specific fidelity checklist.
Sleep Navigator feasibility (Sleep Navigation activities completed among those randomized to receive Sleep Navigation) | within 8 months of baseline assessment
  Feasibility will be measured using data from the caregiver-completed qualitative interview.
Acceptability of the Sleep Navigation program (Treatment Evaluation Inventory-Short Form) | within 8 months of baseline assessment
  Acceptability of the Sleep Navigation program will be measured through the Treatment Evaluation Inventory-Short Form that has been adapted for the Sleep PASS program. This measure is rated on a 5-point Likert scale (1=strongly disagree; 2=disagree; 3=neutral; 4=agree; and 5=strongly agree) with a range in raw score from 11 to 55. Higher total scores indicate better acceptability.
Acceptability of the Sleep Navigation program (Multicultural Therapy Competency Inventory) | within 8 months of baseline assessment
  Sleep Navigation acceptability will be measured through the Multicultural Therapy Competency Inventory- Client Version questionnaire that has been adapted for the Sleep PASS program. This measure is rated on a 5-point Likert scale (1=strongly disagree; 2=disagree; 3=neutral; 4=agree; and 5=strongly agree) with a range in raw score from 5 to 25. Higher total scores indicate better outcomes.

SECONDARY OUTCOMES:
Sleep specialty care referral rates | through study completion, an average of 1 year
  The change in referral rates will be measured through the proportion of patients referred for SDB specialty care of those identified with sleep disordered breathing symptoms based on well visit sleep screener over the study period.
Completion of sleep specialty care referral | through study completion, an average of 1 year
  The change in referral completion for child sleep disordered breathing care will be measured through the proportion of patients randomized to Sleep Navigation who complete their specialty care referral of those referred to specialty care.
Caregiver knowledge of Sleep Disordered Breathing (SDB) | at baseline and within 8 months of baseline assessment
  The magnitude and direction of change in caregiver knowledge of SDB will be measured through the obstructive Sleep Disordered Breathing and Adenotonsillectomy knowledge scale for caregivers. This measure is rated on a dichotomous scale (True/False) with a total raw score range of 0 to 39. Correct answers are summed to attain an overall percentage score representing the degree of knowledge level, with a minimum value of zero and a maximum of 100%. A higher percentage indicates better outcomes.
Child SDB symptoms: Pediatric Sleep Questionnaire | at baseline and within 8 months of baseline assessment
  The magnitude and direction of change in child sleep will be measured through the Pediatric Sleep Questionnaire scores, the most validated questionnaire assessing children's SDB symptoms. This measure is rated on a dichotomous scale ("yes" = 1, "no" = 0, and "don't know"=missing). The result is a proportion that ranges from 0.0 to 1.0. Scores greater than 0.33 are considered positive and suggestive of high risk for a pediatric sleep-related breathing disorder.
Child sleep habits: Brief Child Sleep Questionnaire (BCSQ) | at baseline and within 8 months of baseline assessment
  The magnitude and direction of change in child sleep will be measured through the BCSQ which assesses child sleep habits including sleep time, total sleep duration, night waking, aspects of the sleep environment, etc. The BCSQ uses a nominal scale system. Scores on each subscale and the total score are scaled from 0 to 100. Higher scores denote better sleep quality, more positive perception of child sleep, and parent behaviors that promote healthy and independent sleep.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbances | at baseline and within 8 months of baseline assessment
  The PROMIS Sleep Disturbances survey would measure the magnitude and direction of change in child sleep. This measure is rated on a 5-point Likert scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40. The raw scores are converted to a standardized T-score, with higher scores indicating greater severity of sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment | at baseline and within 8 months of baseline assessment
  The PROMIS Sleep-Related Impairment survey would measure the magnitude and direction of change in child sleep. This measure is rated on a 5-point Likert scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40. The raw scores are converted to a standardized T-score, with higher scores indicating greater severity of sleep-related impairment.
Child sleep practices | at baseline and within 8 months of baseline assessment
  Sleep practices would be assessed using the Patient-Reported Outcomes Measurement Information System Sleep Practices survey. This measure assesses 5 sleep practices: sleep timing, sleep routines and consistency, technology use before bedtime, sleep environment, and the need for parental presence to fall asleep. This measure is rated on a nominal scale and 5-point Likert scale. Scores on each subscale and the total score are scaled from 0 to 100. Higher scores indicate better sleep practices.
Child obstructive sleep apnea symptoms | at baseline and within 8 months of baseline assessment
  The change in child obstructive sleep apnea (OSA) symptoms will be measured through the OSA-18, a validated caregiver-completed questionnaire. This measure is rated on a 7-point Likert scale. Total raw score ranges from 18 to 126. Higher scores indicates worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Williamson, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Archbold KH, Pituch KJ, Panahi P, Chervin RD. Symptoms of sleep disturbances among children at two general pediatric clinics. J Pediatr. 2002 Jan;140(1):97-102. doi: 10.1067/mpd.2002.119990. PMID 11815771
- [Background] Rosen CL, Larkin EK, Kirchner HL, Emancipator JL, Bivins SF, Surovec SA, Martin RJ, Redline S. Prevalence and risk factors for sleep-disordered breathing in 8- to 11-year-old children: association with race and prematurity. J Pediatr. 2003 Apr;142(4):383-9. doi: 10.1067/mpd.2003.28. PMID 12712055
- [Background] Bonuck KA, Chervin RD, Cole TJ, Emond A, Henderson J, Xu L, Freeman K. Prevalence and persistence of sleep disordered breathing symptoms in young children: a 6-year population-based cohort study. Sleep. 2011 Jul 1;34(7):875-84. doi: 10.5665/SLEEP.1118. PMID 21731137
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Boss EF, Smith DF, Ishman SL. Racial/ethnic and socioeconomic disparities in the diagnosis and treatment of sleep-disordered breathing in children. Int J Pediatr Otorhinolaryngol. 2011 Mar;75(3):299-307. doi: 10.1016/j.ijporl.2010.11.006. Epub 2011 Feb 4. PMID 21295865
- [Background] Meltzer LJ, Plaufcan MR, Thomas JH, Mindell JA. Sleep problems and sleep disorders in pediatric primary care: treatment recommendations, persistence, and health care utilization. J Clin Sleep Med. 2014 Apr 15;10(4):421-6. doi: 10.5664/jcsm.3620. PMID 24733988
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077